CLINICAL TRIAL: NCT04800497
Title: Finding The Seeds Of Recurrence: The Role Of The Liquid Biopsy To Detect Circulating Tumor Cells As Markers Of Advanced Disease And Prognosis In HCC
Brief Title: The Role Of Circulating Tumor Cells As Markers Of Advanced Disease And Prognosis In HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); Niguarda Hospital (Other); Humanitas Clinical and Research Center (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Fabrizio Romano, Prof. Fabrizio Romano, University of Milano Bicocca
Other Study IDs: FINDINGBIOREC
Record Dates: First submitted 2021-02-22; First posted 2021-03-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma; Recurrent Hepatocellular Carcinoma; Circulating Tumor Cell
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononucleate cells (PBMC) and liver tissue samples from tumor and peritumoral parenchyma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients resected for hepatocellular carcinoma: Surgical resection, peripheral blood sampling
  Interventions: Procedure: Hepatic resection
- Patients who underwent surgery for benign diseases: Surgical resection, peripheral blood sampling

INTERVENTIONS:
Procedure: Hepatic resection — Hepatic resection for HCC
  Groups: Patients resected for hepatocellular carcinoma

SUMMARY:
Hepatocellular carcinoma (HCC) recurs in up to 60% of patients who undergo resection. Circulating tumor cells (CTC) have been advocated as promotors of the recurrence. However, their role as prognostic markers in the surgical setting is unclear. The aim of the present study has been to assess the association between CTC from peripheral blood samples and the risk of recurrence after surgery.

Patients with a first diagnosis of HCC, no previous treatment for this condition, no other oncological history, and BCLC stage 0-A-B will be enrolled in 2 centers. Patients will undergo to serial liquid biopsies (i.e., a 15ml peripheral blood sample on each time point) at day 0-30-90-180-365 after surgery. After isolation of peripheral blood mononucleate cells, CTC will be detected by FACSymphony™ and subsequently the following markers will be identified: EpCAM, N-cadherin (N-cad) and CD90. Epithelial-mesenchymal transition (EMT) will be analyzed by an index estimated as the ratio between the number of EpCAM+/N-cad- and EpCAM+/N-cad+ cells (EMT Index). Patients will be divided according to the recurrence status.

DETAILED DESCRIPTION:
Liquid biopsy may allow a better stratification of patients according to their estimated prognosis. As well in other tumors (e.g. breast cancer), molecular characterization is permitting not only to better understand the pathological pathways which lead tumorigenesis and progression, but also to drive specific treatments tailored on the specificity of the patient disease. Liquid biopsy is very easy and cheap to perform, since it consist in a simple venous blood sample which will be investigated by cells sorter to identify specific populations of cells.

In hepatocellular carcinoma is common to assist on an elevated recurrence rate: patients who have been treated with a curative intent, in 70% of cases relapse. In these cases, patients often had an underlying inflammatory liver disease, as cirrhosis, which may drive the relapse as an oncogenetic factor. Cirrhosis is a well-know risk factor for developing hepatocellular carcinoma in general. Because of this, in clinical practice is almost difficult to distinguish if the new nodule we have diagnosed should be considered as a real recurrence of the first treated tumor, or a de-novo occurrence linked to the unchanged underlying tumorigenesis boost, which may be effectively cured only after liver transplantation. Several retrospective studies already demonstrated the advantage, in terms of disease-free-survival and overall-survival, of a de-novo occurrence in respect to a real metastatic presentation. However, no one has reached any specific clinical or morphological markers to distinguish between these two conditions. Characterization of the nature of the recurrent nodule has been obtained only by genetic and molecular evaluation of the tumors heterogeneity. Nevertheless, this characterization nowadays is possible only with research intent, and on histological specimen, which could be provided only after an eventual decision of redo-surgery to treat the considered recurrence. Indication on how to treat HCC recurrence after surgery still lacks. Our hypothesis is founded on the "seed and oil" theory, which is basically founded on the evidence of the presence of circulating tumor cells (CTCs) in the blood stream. These cells may be spread from the original tumors as an hallmark of advance cancer, which has already developed the invasiveness characteristic. It is our opinion that tumors in an early stage do not release, or not in the same rate or quality, CTCs in the bloodstream as advanced tumor does. We considered an advanced tumor the one which may has already microvascular invasion and/or satellitosis, which may be the histological signs of an advanced and already systemic stage. Patients with CTCs identified at the liquid biopsy may be associated with a worsen prognosis, accounting for an increased rate of early recurrence and overall recurrence, even in case of transplantation. In addition, the "seed and oil" theory, associated with the "rehoming theory" may justified, from a bio-oncological point of view, the cases of recurrence in the transplant setting, when the whole organ, and the relative oncogenetic risk factors, is treated by substitution. Finally, from a pathophysiological point of view, we want to demonstrate that recurrent intra-hepatic nodules (IM) are due to circulating tumour cells'seeding, permitting a better understanding of carcinogenesis in those tumours.

* Primary objective: to evaluate the association between variation in CTCs - determined in blood samples - and overall survival and disease-free-survival in HCC patients before and after surgery (either resection and transplant).
* Secondary objective: to evaluate if the positive identification of CTCs in blood samples is associated with the intra-hepatic metastatic pattern of recurrence in either resected patients and transplanted one.
* Tertiary objective: to evaluate and to monitor the role of different clinical, biochemical, radiological and histopathological variables in determining the recurrence after surgery and their eventual relationship with the presence and rate of CTCs Patients enrollment will be assessed by the surgical divisions of this study, usually during the outpatient clinic visit before the surgical operation. In that moment patients will be candidate for this study, and, if they accept to participate, researchers will acquire the written consent. Enrolled patients will be codified by an alpha-numeric number to preserve the identity. Researchers who will be employed in the laboratory where the CTCs will be analyzed will not be able to trace the owner of the sample, and they will not have the access to the clinical data (blind analysis).

Before surgery for each patient liquid biopsy from peripheral blood will be collected (in the same time of routine blood analysis). Samples will be used to analyze CTCs rate and type by FACSARIA III (BD bioscience). During surgery, a fresh slice of the tumor and near health liver will be collected by an expert pathologist, who will use section(s) for the usual histological evaluation as provided by the best clinical practice and international guidelines. The remaining sections will be maintained on ice during shipment to the laboratory unit. Researchers will perform alive hepatic cells isolation and storage under sterile conditions. Then, hepatic cells will be analyzed with FACSARIA III and used for further in-vitro experiments.

Liquid biopsy will be performed again at 30th post-operative day during the first outpatient visit, and then every six months, in accordance and in parallel with the local follow-up protocols. Liquid biopsy performed during follow-up will be managed as the pre-operative one, during the normal tests provided for clinical purpose. Follow-up will be closed at 30 months.

All operations will be performed by surgeons with large experience in liver surgery. The resection technique will be at surgeon preference, according to local protocol, good clinical practise and national guidelines. All surgeons adopted the same criteria to select the surgical strategy: baseline variables of liver function, tumour location and diameter, and number of nodules. Restaging Ultrasonography (US) will be performed intra-operatively for each patient. After tumor removal, a pathologist involved in this study will sample the tumor to obtain a fresh-frozen section of the tumor, with the related healthy liver tissue, to store it for further analysis. This sample should be performed in accordance with international guidelines and local ethical agreement, and it must always guarantee the correct material to perform the histological diagnosis. If the tissue removed from the patient enrolled in this study does not allow to perform the sample for the study without affecting the optimal histological diagnosis, the patient will be excluded from the study and no sampling will be executed.

For all patients 20 mL fasting blood sample will be collected in a sterile vacuum tube. The collection will be done in the same time of routine preoperative blood samples or planned follow-up controls, since no others invasive procedure should be provided to patients since their enrollment in the study. The blood sample will be stored at 4°C and handled within 6 hours. Then, 5 mL will be centrifuged at 3000 rpm for 10 minutes at 4°C, the plasma phase will be collected and aliquoted in 1.5 mL sterile tubes and stored at -80°C until use or shipment. Then, we will isolate peripheral blood mononucleate cells (PBMC) through Ficoll gradient from the remaining 15 mL. After isolation, live PBMC will be frozen in standard media 20% Fetal Bovin Serum (FBS) 10% Dymethil Sulfoxide (DMSO) and stored in liquid nitrogen until use.

For all patient liver tissue sample will be collected and tumor (T) portion will be separated from peritumor (PT) portion. From T and PT tissue will be isolated consequentially Human Hepatocytes (HC), Kupffer cells (KC), Liver Sinusoidal Endothelial Cells (LSEC) and Human Stellate Cells (HSC) under sterile conditions. Briefly, liver tissue will be placed in a Petri dish and cut with sterile scalpel. Then, cut liver will be incubated in a 50 mL tube with collagenase P (1mg/mL) at 37°C for 45 minutes. After incubation, collagenase P will be inactivated adding 20% FBS Hank's Balance Salt Solution (HBSS) and cell suspension will be centrifuged 50g 5 minutes at 4°C. The supernatant, containing liver non-parenchymal cells (NPC), will be collected in a new 50 mL tube and pellet will be washed with Phosphate Buffer Solution (PBS). HC and NPC will be frozen in standard media 20% FBS 10% DMSO and stored in liquid nitrogen until use.

A fragment of T and PT will be stored in RNAlater solution at -80°C. For CTC identification PBMC will be thawed, resuspended in standard media and sorted with FACSARIA III (BD bioscience) through EpCAM+, CD47+, CD133+. The percentage of single positive cells (EpCAM+, CD47+ and CD133+) and triple positive cells (EpCAM/CD47/CD133+++) will be evaluated and the total CTC number will be calculated. CTC will be tested for their replicative and invasive capacity. Using cell proliferation and invasion assay we will evaluate CTC doubling time (time needed for the cells to double in number), growth rate (gr=[ln(N(t)/N(0)]/t; N(t)= the number of cells at time t, N(0)= the number of cells at time 0, t= time) and invasion rate.

After CTC characterization we will analyse HC and NPC, using the positive markers previously described, in order to evaluate the exact CTC hepatic derivation.

The biological material will be shipped by expert private transport and stored to the laboratory in "Università degli Studi del Piemonte Orientale".

The recurrence patterns will be evaluated as follow. Local recurrence will be defined as a recurrence on the same liver segment in case of Parenchyma Sparing Resection, or on the surgical hedge of the nearest segments in case of Anatomic Resection. Thus, it will be evaluated the number of recurrent nodules (single versus multiple), the location of recurrence (intrahepatic versus extrahepatic or both), the size of the main recurrent nodule and the liver segment. All this evaluations on recurrence will be made by CT scan or MRI scan during follow-up, as the local follow-up protocols provide.

All the patients will be followed using a local protocol including measurement of serum α-FP, total bilirubin, GGT, ALP, Albumine, INR, blood count, electrolyte count, ultrasound, contrast Computed Tomography (CT) or magnetic Resonance Imaging (MRI) and office visits. Patients usually are checked every 3 months during the first postoperative year and every 6 months thereafter. When the recurrence occurred, the cases are discussed in a multidisciplinary setting, involving radiologist, hepatologist, surgeon, interventional radiologist, radiotherapist and oncologist. Overall-Survival (OS) is defined as time interval (in months) from surgery to patient death. Data will be censored in case of loosed patient at the follow-up screening. Disease-Free Survival (DFS) is defined as time interval (in months) from surgery to recurrence or death. In case of no recurrence, data will be censored at the date of the last available follow-up. Tumor-Specific-Survival (TSS) is defined as the time interval in months between surgery and tumor-related death.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocarcinoma diagnosis confirmed by radiology and committed to surgery (resection or OLT) with curative intent.
* First diagnosis and first treatment of hepatocellular carcinoma.
* BCLC 0 - A - B
* Histological confirmation of hepatocarcinoma at the histological specimen.
* Availability of a fresh frozen section of the tumor obtained during the surgical procedures

Exclusion Criteria:

* Other tumors in the clinical history.
* Presence of autoimmune liver diseases (eg. sclerotising cholangitis, primary biliary cirrhosis etc.).
* Patients treated with surgery in case of not-curative intent (palliation, best supportive care, etc).
* Histopathological specimen of combined liver primary neoplasms (e.g. 'epatocolangiocarcinoma').
* Patients previously treated for HCC with other therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned number of subjects to be screened for resection group: almost 40 per year (patients treated/year in centres already registered as participating). Final number of enrolled at the end of the period: 80 patients. Planned number of subjects to be screened for OLT group: almost 30 per year. Final number of enrolled at the end of the period: 60 patients.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Association between circulating tumor cells and disease-free-survival | 5 years
  To evaluate the association between variation in CTCs - determined in blood samples - and disease-free-survival in HCC patients after surgery.

SECONDARY OUTCOMES:
Association between circulating tumor cells and overall survival | 5 years
  To evaluate the association between variation in CTCs - determined in blood samples - and overall survival in HCC patients after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Romano, Principal Investigator — University of Milano Bicocca
Locations (4):
- Italy (4):
  - Ospedale San Gerardo, Monza, MB
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Università del Piemonte Orientale, Novara
  - Humanitas Research Hospital, Rozzano

IPD SHARING:
Plan to Share IPD: Undecided